CLINICAL TRIAL: NCT00306878
Title: Phase I Study of BMS-188667 (CTLA4Ig) in Patients With Psoriasis Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM101-001
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Abatacept

INTERVENTIONS:
Drug: Abatacept

SUMMARY:
The purpose of this clinical research study is to determine the safety, pharmacokinetics, immunogenicity in humans, the recovery time required from the biologic effects and the optimal biologic dose range of BMS188667 (CTLA4Ig)

ELIGIBILITY:
Inclusion Criteria:

* Men or women who received adequate counseling and were judged reliabel in their use of contraceptive measures.
* Diagnosis and documentation of stable psoriasis vulgaris of at least 6 months duration.
* Psoriasis vulgaris total body surface area involvement between 10% and 49% (Overall Disease Severity Score [ODSS]of 4-7 inclusive).
* Failure of toxicity or inefficacy of at least one standard antipsoriatic therapy including topical treatment, etretinate, phototherapy, or methotrexate.

Exclusion Criteria:

* Treatment with: a) Retinoids within 2 years, b) cyclosporin A, systemic corticosteroids, methotrexate, or an investigational agent within 16 weeks, c) any phototherapy or photochemotherapy within 4 weeks d) any topical psoriasis treatment other than emollients within 2 weeks prior to enrollment.
* No clinical response to a prior adequate therapeutic trial of cyclosporin A
* Prolonged exposure to the sun within 4 weeks prior to the first dose.
* Guttate, erythrodermic, or pustular psoriasis.
* Spontaneously improving or rapidly deteriorating psoriasis vulgaris.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45
Dates: Start 1995-08; Primary Completion 1997-05 (Actual); Study Completion 1997-05 (Actual)

PRIMARY OUTCOMES:
Change relative to pretreatment of the Overall Disease Severity Score (ODSS) for psoriasis vulgaris as assess by a blinded observer. Phage-Neutralizing anitbody titer | at Day 43

SECONDARY OUTCOMES:
Physician's globas Assessment | at Day 36
Phage-neutralizing antibody titer | at Day 16 and Day 29
Mean percentage of anti-bacteriophage FX174 antibody of IgG isotype in sera collected | at Day 43

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Local Institution, Boston, Massachusetts
  - Local Institution, Ann Arbor, Michigan
  - Local Institution, New York, New York
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania